CLINICAL TRIAL: NCT00736918
Title: A Randomized Controlled Multicenter Trial of Post-Suicide Attempt Case Management for the Prevention of Further Attempts in Japan (ACTION-J)
Brief Title: RCT of Post-Suicide Attempt Case Management (ACTION-J)
Acronym: ACTION-J
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Foundation for Neuroscience and Mental Health (Other)
Collaborators: National Center of Neurology and Psychiatry, Japan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: J-MISP-01; C000000444 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Suicide Attempt
Keywords: Suicide Attempt
MeSH Terms: conditions — Suicide, Attempted | interventions — Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Case management (Experimental): Case management
  Interventions: Behavioral: Case management
- Enhanced usual care (Active Comparator): Enhanced usual care
  Interventions: Other: Enhanced usual care

INTERVENTIONS:
Behavioral: Case management — Case management, Usual clinical practice and Providing paper based information for suicide prevention
  Arms: Case management
Other: Enhanced usual care — Usual clinical practice and Providing paper based information for suicide prevention
  Arms: Enhanced usual care

SUMMARY:
This study will determine the effectiveness of continuous follow-up care by case manager in preventing further suicide attempts

DETAILED DESCRIPTION:
It is well known that many subjects who survived a suicide attempt will make further suicide attempts, even after the medical treatment at critical emergency unit. To examine the effectiveness of continuous follow-up care by case manager after the suicide attempt, a randomized, controlled, multicenter trial by J-MISP (Japanese Multimodal Intervention Trials).This research project is one of the strategic research projects funded by The Japanese Ministry of Health, Labor and Welfare. In this study, J-MISP will implement the intervention for suicide attempters, a considerably high-risk group of further suicide attempts, who are transported by emergency services.

ELIGIBILITY:
Inclusion Criteria:

1. Over 20 years old
2. Suffering from Axis I disorder
3. Had intent for suicide (confirmed more than 2 times)
4. Able to understand this study and provide informed consent
5. Able to have interview before trial registry and psycho education at hospital
6. Able to have interview for assessment at continuous follow-up care by case manager at the hospital

Exclusion Criteria:

1. Not suffering from Axis I disorder as a primary diagnosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 914 (Actual)
Dates: Start 2006-06; Primary Completion 2011-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
First recurrent suicide behavior (suicide attempted and completed suicide) | Minimum 1.5 year

SECONDARY OUTCOMES:
Any cause of death | Minimum 1.5 year
Repeated recurrent incidence of suicide attempts | Minimum 1.5 year
Utilization or personal or social resources | Minimum 1.5 year
Number of self-injury | Minimum 1.5 year
Health care utilization | Minimum 1.5 year
Physical function | Minimum 1.5 year
Beck hopeless scale | Minimum 1.5 year
SF-36 | Minimum 1.5 year
Adverse events | Minimum 1.5 year

OTHER OUTCOMES:
Incidence proportion of the first episode of recurrent suicidal behaviour (attempted suicide or completed suicide) | at 1 month after the randomization
Incidence proportion of the first episode of recurrent suicidal behaviour (attempted suicide or completed suicide) | at 3 months after the randomization
Incidence proportion of the first episode of recurrent suicidal behaviour (attempted suicide or completed suicide) | at 6 months after the randomization
Incidence proportion of the first episode of recurrent suicidal behaviour (attempted suicide or completed suicide) | at 12 months after the randomization
Incidence proportion of the first episode of recurrent suicidal behaviour (attempted suicide or completed suicide) | at 18 months after the randomization

CONTACTS AND LOCATIONS:
Overall Officials: Yoshio Hirayasu, MD,PhD, Principal Investigator — Yokohama City University
Locations (18):
- Japan (18):
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - National Hospital Organization, Mito Medical Center, Mito, Ibaraki
  - Tsuchiura Kyodo Hospital, Tsuchiura, Ibaraki
  - Tsukuba Medical Center, Tsukuba, Ibaraki
  - Iwate Medical University Hospital, Morioka, Iwate
  - Kitazato University Hospital, Sagamihara, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Nara Medical University Hospital, Kashihara, Nara
  - Oita Kouseiren Tsurumi Hospital, Beppu, Oita Prefecture
  - Oita University Hospital, Yufu, Oita Prefecture
  - Kansai Medical University Takii Hospital, Moriguchi, Osaka
  - National Hospital Organization, Osaka Medical Center, Osaka, Osaka
  - Kinki University Hospital, Sayama, Osaka
  - Saitama Medical University Medical Center, Kawagoe, Saitama
  - Saitama Medical University Hospital, Morohongō, Saitama
  - Nihon Medical University Hospital, Tokyo, Tokyo
  - Showa University Hospital, Tokyo, Tokyo

REFERENCES:
- [Background] Hirayasu Y, Kawanishi C, Yonemoto N, Ishizuka N, Okubo Y, Sakai A, Kishimoto T, Miyaoka H, Otsuka K, Kamijo Y, Matsuoka Y, Aruga T. A randomized controlled multicenter trial of post-suicide attempt case management for the prevention of further attempts in Japan (ACTION-J). BMC Public Health. 2009 Sep 26;9:364. doi: 10.1186/1471-2458-9-364. PMID 19781096
- [Background] Kawanishi C, Hirayasu Y, Ariga T, Ishizuka N, Yamada M, Takahashi K. ["ACTION-J", a multi-center joint study for the development of strategies to prevent recurrence of suicidal ideation (a strategic study for anti-suicide policies supported by the Health, Labor and Welfare Ministry): its background and research outline]. Seishin Shinkeigaku Zasshi. 2008;110(3):230-7. No abstract available. Japanese. PMID 18524048
- [Derived] Inui-Yukawa M, Miyaoka H, Yamamoto K, Kamijo Y, Takai M, Yonemoto N, Kawanishi C, Otsuka K, Tachikawa H, Hirayasu Y. Effectiveness of assertive case management for patients with suicidal intent. Psychiatry Res. 2021 Oct;304:114125. doi: 10.1016/j.psychres.2021.114125. Epub 2021 Jul 19. PMID 34332432
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Kawanishi C, Aruga T, Ishizuka N, Yonemoto N, Otsuka K, Kamijo Y, Okubo Y, Ikeshita K, Sakai A, Miyaoka H, Hitomi Y, Iwakuma A, Kinoshita T, Akiyoshi J, Horikawa N, Hirotsune H, Eto N, Iwata N, Kohno M, Iwanami A, Mimura M, Asada T, Hirayasu Y; ACTION-J Group. Assertive case management versus enhanced usual care for people with mental health problems who had attempted suicide and were admitted to hospital emergency departments in Japan (ACTION-J): a multicentre, randomised controlled trial. Lancet Psychiatry. 2014 Aug;1(3):193-201. doi: 10.1016/S2215-0366(14)70259-7. Epub 2014 Aug 5. PMID 26360731